CLINICAL TRIAL: NCT03334253
Title: Low-Dose Atropine for Treatment of Myopia (Myopia Treatment Study)
Brief Title: Low-Dose Atropine for Treatment of Myopia
Acronym: MTS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTS1; 2U10EY011751 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Myopia
Keywords: Myopia; atropine
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: The current study is designed as an efficacy study, making effort to maximize adherence to treatment group assignments. After a run-in phase during which all participants are treated with daily artificial tear eyedrops for 2-4 weeks (and glasses are updated if required) to assess their ability to adhere to daily eye drops, participants are randomly assigned to daily atropine or placebo for 24 months, followed by 6 months off treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Cycloplegic autorefraction, axial length, and additional biometry will be measured by a masked examiner at all follow-up visits using the same instrumentation on the participant throughout the study. Masking will be accomplished by having site personnel administer cyclopentolate to both eyes of each participant and wait 30 minutes before he/she sees the masked examiner. The masked examiner may be a technician or an investigator and must be certified to complete these measurements. Parents, patients, and investigators are also masked to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atropine Group (Experimental): 0.01% atropine eyedrops administered 1 drop to each eye daily in each eye for 24 months, followed by 6 months off atropine eyedrops
  Interventions: Drug: Atropine
- Placebo Group (Placebo Comparator): Placebo eyedrops administered 1 drop to each eye daily in each eye for 24 months, followed by 6 months off placebo eyedrops
  Interventions: Other: Placebo Eyedrops

INTERVENTIONS:
Drug: Atropine — Daily 0.01% atropine eyedrops
  Other Names: Low-Dose Atropine
  Arms: Atropine Group
Other: Placebo Eyedrops — Daily placebo eyedrops
  Arms: Placebo Group

SUMMARY:
Study Objectives

The objectives for this randomized trial are:

1. To determine the efficacy of daily low-dose atropine (0.01%) for slowing myopia progression over a two-year treatment period in children aged 5 to less than 13 years (Primary Outcome On-Treatment).
2. To determine the efficacy of atropine treatment on myopia progression 6 months following cessation of low-dose atropine treatment (Secondary Outcome Off-Treatment).

Synopsis of Study Design The current study is designed as an efficacy study, making effort to maximize adherence to treatment group assignments. After a run-in phase during which all participants are treated with daily artificial tear eyedrops for 2-4 weeks (and glasses are updated if required) to assess their ability to adhere to daily eye drops, participants are randomly assigned to daily atropine or placebo for 24 months, followed by 6 months off treatment.

DETAILED DESCRIPTION:
Study Objectives

The objectives for this randomized trial are:

1. To determine the efficacy of daily low-dose atropine (0.01%) for slowing myopia progression over a two-year treatment period in children aged 5 to less than 13 years with myopia -1.00 to -6.00D at the time of enrollment (Primary Outcome On-Treatment).
2. To determine the efficacy of atropine treatment on myopia progression 6 months following cessation of low-dose atropine treatment (Secondary Outcome Off-Treatment).

Synopsis of Study Design The current study is designed as an efficacy study, making effort to maximize adherence to treatment group assignments. After a run-in phase during which all participants are treated with daily artificial tear eyedrops for 2-4 weeks (and glasses are updated if required) to assess their ability to adhere to daily eye drops, participants are randomly assigned to daily atropine or placebo for 24 months, followed by 6 months off treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years to <13 years at time of enrollment. Children within 4 weeks of their 13th birthday are not eligible.
* Refractive error meeting the following by cycloplegic autorefraction:

  * Myopia -1.00D to -6.00D spherical equivalent (SE) in both eyes
  * Astigmatism <=1.50D in both eyes
  * Anisometropia <1.00D SE
* Gestational age ≥ 32 weeks.
* Birth weight >1500g.
* Parent understands the protocol and is willing to accept randomization to atropine or placebo.
* Is willing to participate in a 2 to 4 week run-in phase using daily artificial tear eyedrops.
* Able to return in 2 to 4 weeks for possible randomization.
* Parent has a phone (or access to phone) and is willing to be contacted by Investigator's site staff.
* Relocation outside of the area of an active PEDIG site within next 32 months is not anticipated.

Exclusion Criteria:

* Current or previous myopia treatment with atropine, pirenzepine or other anti-muscarinic agent.
* Current or previous use of bifocals, progressive-addition lenses, or multi-focal contact lenses.
* Current or previous use of orthoK, rigid gas permeable, or other contact lenses being used to reduce myopia progression.
* Known atropine allergy.
* Abnormality of the cornea, lens, central retina, iris or ciliary body.
* Current or prior history of manifest strabismus, amblyopia, or nystagmus.
* Prior eyelid, strabismus, intraocular, or refractive surgery.
* Down syndrome or cerebral palsy.
* Females who are pregnant, lactating, or intending to become pregnant within the next 30 months.

  * A negative urine pregnancy test will be required for all females who have experienced menarche.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, MD, MBA, Study Chair — Wilmer Eye Institute; Katherine K Weise, OD, MBA, Study Chair — University of Alabama Birmingham Pediatric Eye Care, Birmingham Health Care
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Emory Eye Center Dept of Ophthalmology, Atlanta, Georgia
  - St Luke's Hospital, Boise, Idaho
  - Illinois College of Optometry, Chicago, Illinois
  - Ticho Eye Associates, Chicago Ridge, Illinois
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - Eye Care Associates, Inc., Poland, Ohio
  - Dean A. McGee Eye Institute, University of Oklahoma, Oklahoma City, Oklahoma
  - Casey Eye Institute, Portland, Oregon
  - Vanderbilt University Medical Center - Vanderbilt Eye Institute, Nashville, Tennessee
  - University of Houston College of Optometry, Houston, Texas
  - Rocky Mountain Eye Care Associates, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the protocol and publication of the primary manuscript, the data will be made available for the duration of the grant and any future grants.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Result] Repka MX, Weise KK, Chandler DL, Wu R, Melia BM, Manny RE, Kehler LAF, Jordan CO, Raghuram A, Summers AI, Lee KA, Petersen DB, Erzurum SA, Pang Y, Lenhart PD, Ticho BH, Beck RW, Kraker RT, Holmes JM, Cotter SA; Pediatric Eye Disease Investigator Group. Low-Dose 0.01% Atropine Eye Drops vs Placebo for Myopia Control: A Randomized Clinical Trial. JAMA Ophthalmol. 2023 Aug 1;141(8):756-765. doi: 10.1001/jamaophthalmol.2023.2855. PMID 37440213
- [Derived] Weise KK, Repka MX, Zhu Y, Manny RE, Raghuram A, Chandler DL, Summers AI, Lee KA, Kehler LAF, Pang Y, Allen MS, Anderson HA, Erzurum SA, Golden RP, Koutnik CA, Kuo AF, Lenhart PD, Mokka PL, Petersen DB, Ticho BH, Wiecek EK, Yin H, Beaulieu WT, Kraker RT, Holmes JM, Cotter SA; Pediatric Eye Disease Investigator Group. Baseline factors associated with myopia progression and axial elongation over 30 months in children 5 to 12 years of age. Optom Vis Sci. 2024 Oct 1;101(10):619-626. doi: 10.1097/OPX.0000000000002187. PMID 39480129

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred patients were enrolled into the run-in phase; 13 were ineligible for randomization
Period: Overall Study
Arm/Group | Atropine Group | Placebo Group
Started | 125 | 62
Completed | 118 | 57
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Moved residence | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atropine Group | Placebo Group | Total
Number analyzed (Participants) | 125 | 62 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.8) | 10.1 (1.8) | 10.1 (1.8)
Age, Customized [Count of Participants; unit: Participants]
  5 to <7 years | 6 | 3 | 9
  7 to <9 years | 28 | 13 | 41
  9 to <11 years | 50 | 20 | 70
  11 to <13 years | 41 | 26 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 36 | 101
  Male | 60 | 26 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (not Hispanic or Latino) | 58 | 28 | 86
  White Hispanic or Latino | 21 | 9 | 30
  Black | 20 | 14 | 34
  East Asian | 16 | 4 | 20
  West Asian / South Asian | 4 | 2 | 6
  More Than one race | 6 | 5 | 11
Eye Color [Count of Participants; unit: Participants]
  Brown | 82 | 41 | 123
  Not Brown | 43 | 21 | 64
Number of Biological Parents with Myopia [Count of Participants; unit: Participants]
  0 | 16 | 11 | 27
  1 | 51 | 24 | 75
  2 | 52 | 20 | 72
  Myopia history unknown for one or both parents | 6 | 7 | 13
Current Refractive Correction (Single-vision Spectacles or Contact Lenses) [Count of Participants; unit: Participants]
  Yes | 125 | 61 | 186
  No | 0 | 1 | 1
Distance Visual Acuity in Habitual Refractive Correction (Mean of Both Eyes) [Count of Participants; unit: Participants]
  <-0.2 logMAR | 0 | 1 | 1
  -0.2 to < -0.1 logMAR | 18 | 5 | 23
  -0.1 to < 0.0 logMAR | 62 | 35 | 97
  0.0 to < 0.1 logMAR | 36 | 16 | 52
  0.1 to < 0.2 logMAR | 9 | 5 | 14
Mean OD and OS Flat Corneal Radius [Mean (Standard Deviation); unit: Diopters squared] — Population: Flat corneal radius was not available for 1 patient in the placebo group.
  Diopters squared
    number analyzed (Participants) | 125 | 61 | 186
    (all) | 43.4 (1.4) | 43.6 (1.4) | 43.4 (1.4)
Mean OD and OS Anterior Chamber Depth [Mean (Standard Deviation); unit: millimeter] | 3.8 (0.2) | 3.9 (0.2) | 3.9 (0.2)
Mean OD and OS Lens Thickness [Mean (Standard Deviation); unit: millimeters cubed] — Population: Lens thickness was not available for some patients (N=53 in atropine and N=27 in placebo) because the biometer used did not provide a lens thickness reading due to measurement difficulty.
  millimeters cubed
    number analyzed (Participants) | 72 | 35 | 107
    (all) | 3.4 (0.2) | 3.3 (0.2) | 3.3 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Group Comparison of Change in Spherical Equivalent Refractive Error.
Description: The primary analysis will be a treatment group comparison of change from baseline to 24-months in spherical equivalent refractive error (SER), as measured by a masked examiner using cycloplegic autorefraction (on-treatment comparison).
  The mean of the three readings from autorefraction in each eye will be calculated and then the mean of both eyes for each participant will be used for the analysis.
  The treatment group difference (atropine - placebo) and a 95% confidence interval will be calculated based on the model estimates at 24 months.
Time Frame: At 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atropine Group | Placebo Group
Number analyzed (Participants) | 119 | 58
Participants
  <=-3.50 Diopters | 0 | 0
  >-3.50 to -3.00 Diopters | 1 | 0
  >-3.00 to -2.50 Diopters | 1 | 0
  >-2.50 to -2.00 Diopters | 5 | 2
  >-2.00 to -1.50 Diopters | 8 | 7
  >-1.50 to -1.00 Diopters | 19 | 9
  >-1.00 to -0.50 Diopters | 37 | 18
  >-0.50 to 0.00 Diopters | 46 | 18
  >0 Diopters | 2 | 4
Statistical Analysis 1: Comparison: Atropine Group vs Placebo Group; Null Hypothesis: no difference in mean change in SER from baseline to 24 months between the atropine and placebo groups; Test type: Superiority — The following assumptions were used in the power calculation: * 2:1 randomization * treatment group difference of 0.50D * standard deviation of 0.80D * type 1 error of 5% (2-sided) * up to 10% loss to follow up; Adjusted mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.15] — Atropine - Placebo Adjusted mean difference, adjusting for baseline refractive error, age, iris color (brown vs. not brown), and race (East Asian vs. non-East Asian)

2. Secondary Outcome: Treatment Group Comparison of Change From Baseline to 30 Months in Spherical Equivalent
Description: Treatment group comparison of change from baseline to 30 months in spherical equivalent in each eye as measured by a masked examiner using cycloplegic autorefraction (off-treatment comparison). Calculated based on the model estimates at 24 months.
Time Frame: At 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atropine Group | Placebo Group
Number analyzed (Participants) | 118 | 57
Participants
  <=-3.50 Diopters | 1 | 0
  >-3.50 to -3.00 Diopters | 2 | 1
  >-3.00 to -2.50 Diopters | 5 | 0
  >-2.50 to -2.00 Diopters | 5 | 3
  >-2.00 to -1.50 Diopters | 8 | 6
  >-1.50 to -1.00 Diopters | 22 | 11
  >-1.00 to -0.50 Diopters | 35 | 20
  >-0.50 to 0.00 Diopters | 36 | 13
  >0 Diopters | 4 | 3
Statistical Analysis 1: Comparison: Atropine Group vs Placebo Group; Null Hypothesis: no difference in mean change in SER from baseline to 24 months between the atropine and placebo groups; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.04, 95% CI 2-sided [-0.25 to 0.17] — Atropine-Placebo Adjusted mean difference, adjusting for baseline refractive error, age, iris color (brown vs. not brown), and race (East Asian vs. non-East Asian)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study, baseline to 30 months.
Arm/Group | Atropine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/125 | 0/62
Other Adverse Events (participants affected / at risk) | 109/125 | 56/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atropine Group (N=125) | Placebo Group (N=62)
Hospitalization (General disorders) | 2 (2) | 0 (0) — Hospitalization for issues unrelated to the study, two hospitalizations include: one participant undergoing hip surgery for a pre-existing condition; one participant hospitalized for COVID-19.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atropine Group (N=125) | Placebo Group (N=62)
Eye Irritiation (Eye disorders) | 90 | 51
Photophobia (Eye disorders) | 32 | 17
Vision Blurred (Eye disorders) | 17 | 10
Allergic Conjunctivitis (Eye disorders) | 10 | 5
Ocular Discomfort (Eye disorders) | 8 | 5
Visual Impairment (Eye disorders) | 6 | 2
Blepharitis (Eye disorders) | 6 | 1
Meibomian gland dysfunction (Eye disorders) | 3 | 3
Eye Pain (Eye disorders) | 9 | 0
Dry Eye (Eye disorders) | 3 | 1
Hordeolum (Eye disorders) | 2 | 2
Accommodation Disorder (Eye disorders) | 3 | 0
Optic Disc Drusen (Eye disorders) | 1 | 0
Headache (Eye disorders) | 1 | 0
Visual Acuity Reduced (Eye disorders) | 2 | 0
Vitreous Floaters (Eye disorders) | 2 | 0
Eye injury (Eye disorders) | 0 | 2
Ocular hyperaemia (Eye disorders) | 2 | 0
Retinal degeneration (Eye disorders) | 2 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Foreign body in eye (Eye disorders) | 0 | 1
Meibomianitis (Eye disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Dermatitis contact (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Pruritus (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Chalazion (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 1 | 0
Corneal Scar (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT03334253/Prot_001.pdf
  • Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03334253/SAP_002.pdf
  • Informed Consent Form (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03334253/ICF_000.pdf